CLINICAL TRIAL: NCT03654404
Title: A Proof-of-Concept Trial of a Positive Psychology Intervention for Allogeneic Stem Cell Transplant Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: Harvard Medical School (HMS and HSDM) (Other)
Responsible Party: Principal Investigator, Hermioni L.Amonoo, MD, MPP, MPH, Director, Well-Being and Cancer Research Program, Brigham and Women's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 18-225
Record Dates: First submitted 2018-08-29; First posted 2018-08-31 (Actual); Results first posted 2022-01-19 (Actual); Last update posted 2024-06-12 (Actual); Status verified 2024-05

CONDITIONS: Hematologic Malignancy; Hematopoietic/Lymphoid Cancer; Blood Cancer
Keywords: Hematopoietic Stem Cell Transplant; Positive Psychology; Hematologic malignancy; Positive Psychological Intervention
MeSH Terms: conditions — Hematologic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Positive Psychology (Experimental): Participants will receive check-in/psychosocial support phone calls at weeks four, eight and twelve following enrollment.
  At approximately 100-days post-HSCT, participants will begin an 8-week positive-psychology program involving weekly calls with an interventionist, in this case the principal investigator, and exercises (i.e. writing a letter of gratitude, identifying personal strengths, planning meaningful and enjoyable activities).
  Participants will complete self-assessment questionnaires to measure positive affect, health behaviors, and overall function before and after completing the Positive Psychology Intervention.
  Interventions: Behavioral: Positive Psychology Intervention

INTERVENTIONS:
Behavioral: Positive Psychology Intervention — Weekly phone calls with the study interventionist and positive psychology exercises over an 8-week period. The positive psychology program exercises includes three modules: gratitude-based activities, strength-based activities, and meaning-based activities.

SUMMARY:
The goal of this research study is to find out if a novel phone-based positive psychology intervention that focuses on improving health behaviors and positive emotions can help improve mood, health related quality of life, and overall function in patients who have just undergone hematopoietic stem cell transplantation as part of blood cancer treatment.

DETAILED DESCRIPTION:
Hematopoietic stem cell transplantation (HSCT) is a rigorous treatment for blood cancer patients that can be life-saving, but often causes psychological distress. The investigators hope that this study will help the research team to develop and implement a positive psychological intervention designed to help HSCT patients increase positive emotions such as hope, gratitude, and fulfillment while recovering from a stem cell transplant. Participants will be selected after receiving an allogeneic hematopoietic stem cell transplant treatment in the past 30 days at the Dana-Farber Cancer Institute (DFCI).

In this project, the investigators hope to:

1. Test the feasibility and acceptability of a novel, 8-week, phone-based positive psychology intervention in a small cohort of post-HSCT patients (N = 20).
2. Explore potential benefits of completing the intervention on outcomes of interest, such as positive affect and overall function.

Baseline information about enrolled participants will be obtained from patients from the electronic medical record as required for characterization of our population. This information will include data regarding medical history, current medical variables, medications, and sociodemographic data.

Participants will be approached upon nearing their discharge from the hospital, approximately 30 days after their transplant. Between the time of their discharge and their 100-day post-transplant visit, there will be three check-in/psychosocial support phone calls at weeks 4, 8, and 12 after discharge to build rapport and discuss their recovery. Then, at week 14, participants will meet with the principal investigator to complete self-assessment questionnaires. The participants will then complete an 8-week phone-based positive psychology intervention, at the end of which the self-assessment questionnaires will be repeated.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with hematologic malignancies hospitalized for allogeneic HSCT at the DFCI inpatient units who are medically stable and appropriate for study approach
* Ability to speak, read and write English
* Access to a telephone

Exclusion Criteria:

* Current major depressive episode, bipolar disorder, psychosis or active substance use disorder diagnosed via the Mini International Neuropsychiatric Interview (MINI)
* Cognitive deficits impeding a study participant's ability to provide informed consent or participate adequately in the study assessed via the Brief Interview for Mental Status (BIMS)
* Medical conditions precluding interviews

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2018-09-11 (Actual); Primary Completion 2021-03-31 (Actual); Study Completion 2021-07-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hermioni Amonoo, MD, MPP, MPH, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Dana Farber Cancer Institute, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Positive Psychology: Participants will receive check-in/psychosocial support phone calls at weeks four, eight and twelve following enrollment.
  At approximately 100-days post-HSCT, participants will begin an 8-week positive-psychology program involving weekly calls with an interventionist, in this case the principal investigator, and exercises (i.e. writing a letter of gratitude, identifying personal strengths, planning meaningful and enjoyable activities).
  Participants will complete self-assessment questionnaires to measure positive affect, health behaviors, and overall function before and after completing the Positive Psychology Intervention.
  Positive Psychology Intervention: Weekly phone calls with the study interventionist and positive psychology exercises over an 8-week period. The positive psychology program exercises includes three modules: gratitude-based activities, strength-based activities, and meaning-based activities.
Period: Overall Study
Arm/Group | Positive Psychology
Started | 20
Completed | 12
Not Completed | 8
Not completed — Death | 1
Not completed — Lost to Follow-up | 2
Not completed — Withdrawal by Subject | 5

BASELINE CHARACTERISTICS:
Arm/Group | Positive Psychology
Number analyzed (Participants) | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 19
  >=65 years | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.6 (12.78)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 20
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 20
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 20
Optimism [Mean (Standard Deviation); unit: units on a scale] — Optimism was measured using the Life Orientation Test-Revised (LOT-R), a 10-item measure of dispositional (trait) optimism (range 0-24); higher scores indicate greater optimism
  units on a scale | 21.7 (5.1)

OUTCOME MEASURES:

1. Primary Outcome: Feasibility of Positive Psychology (PP) Intervention
Description: Feasibility will be measured by examining the number of completed exercises.
Time Frame: Baseline - week 8 of intervention
Measure: Mean (Standard Deviation); unit: sessions completed out of 8 sessions
Arm/Group | Positive Psychology
Number analyzed (Participants) | 20
sessions completed out of 8 sessions | 8.0 (0)

2. Primary Outcome: Acceptability of Exercises: Ease Score
Description: Participants will provide ratings of ease of completion after each PP exercise, measured on a 10-point Likert scale (score range: 0-10, 0 = very difficult and 10 = very easy). Ratings from all 8 weeks were averaged.
Time Frame: Baseline - week 8 of intervention
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Positive Psychology
Number analyzed (Participants) | 20
score on a scale | 8.0 (2.7)

3. Primary Outcome: Acceptability of Exercises: Utility Score
Description: Participants will provide ratings of utility of completion after each PP exercise, measured on a 10-point Likert scale (score range: 0-10, 0 = not helpful and 10 = very helpful). Ratings from all 8 weeks were averaged.
Time Frame: Baseline - week 8 of intervention
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Positive Psychology
Number analyzed (Participants) | 20
score on a scale | 8.4 (1.9)

4. Secondary Outcome: Changes in PANAS Scores
Description: The positive affect items on the Positive and Negative Affect Schedule (PANAS), a well-validated scale used in other intervention trials and in patients with medical illness, will be used to measure positive affect (Range: 10-50). Higher scores indicate higher levels of positive affect.
Time Frame: Change in score from baseline to 8 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Positive Psychology
Number analyzed (Participants) | 20
score on a scale
  Baseline | 35.17 (5.67)
  Week 8 | 37.08 (4.10)

5. Secondary Outcome: Changes in LOT-R Scores
Description: Life Orientation Test-Revised (LOT-R) is a well-validated 6-item instrument used to measure dispositional optimism (Range: 0-24). Higher scores indicate higher levels of dispositional optimism.
Time Frame: Change in score from baseline to 8 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Positive Psychology
Number analyzed (Participants) | 20
score on a scale
  Baseline | 18.75 (3.98)
  Week 8 | 19.50 (3.55)

6. Secondary Outcome: Changes in HADS Scores
Description: The Hospital Anxiety and Depression Scale (HADS), which consists of the HADS-depression subscale and HADS-anxiety subscale, is a well-validated scale with few somatic symptom items that can confound mood/anxiety assessment in medically ill patients before and after the PP intervention. Both subscales consist of 7 items, and each item is scored on a 0-3 scale, 0 indicating no clinical severity or a lack of symptoms, and 3 indicating significant clinical severity or increased symptom frequency; the maximum score is for each scale 21 and the minimum score is a 0. Higher scores indicate higher levels of depression or anxiety.
Time Frame: Change in score from baseline to 8 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Positive Psychology
Number analyzed (Participants) | 20
score on a scale
  HADS-D Baseline | 6.58 (2.15)
  HADS-D Week 8 | 6.00 (2.00)
  HADS-A Baseline | 5.75 (2.73)
  HADS-A Week 8 | 5.08 (3.20)

7. Secondary Outcome: Changes in FACT-BMT Scores
Description: The Functional Assessment of Cancer Therapy - Bone Marrow Transplant is a 47-item measure of the quality of life in patients undergoing bone marrow transplants before and after the PP intervention. There are five subscales, each including 7 items and various score ranges: Physical Well-Being (0-28), Social/Family Well-Being (0-28), Emotional Well-Being (0-24), Functional Well-Being (0-28), and Transplant (0-40). Each item is scored on a 5-point Likert scale based on patient agreement with each statement: 0 for "not at all," 1 for "a little bit," 2 for "somewhat," 3 for "quite a bit," and 4 for "very much." In each subscale, add items together to get the sum, then the sum is multiplied by 7, and finally, the sum is divided by the number of items answered to obtain the subscale score. The Physical and Emotional subscales are reverse scored. The total score is the sum of the subscale total added together and ranges from 0-148. The higher the score, the better the quality of life.
Time Frame: Change in score from baseline to 8 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Positive Psychology
Number analyzed (Participants) | 20
score on a scale
  Baseline | 107.91 (15.31)
  Week 8 | 110 (18.31)

8. Secondary Outcome: Changes in PROMIS-PF-20 Scores
Description: The Patient-Reported Outcomes Measurement Information System - Physical Function is a well-validated scale used to measure overall function before and after the PP intervention. The PROMIS-Fatigue is scored on a 5-point Likert scale based on how much the person filling out the questionnaire agrees with the statement or question. The minimum value is 1 indicating "not at all" and the maximum value is 5 indicating "very much". Higher scores indicate higher levels of fatigue. The PROMIS-PF scores range from 20-100, with 20 indicating lower or limited levels of physical functioning and 100 indicating no difficulty or higher levels of physical functioning.
Time Frame: Change in score from baseline to 8 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Positive Psychology
Number analyzed (Participants) | 20
score on a scale
  Baseline | 85.67 (8.13)
  Week 8 | 86.33 (10.40)

9. Secondary Outcome: Immediate Impact of Exercises: Optimism Score
Description: Participants will provide ratings of their present level of optimism after each PP exercise, measured on a 10-point Likert scale (score range: 0-10, 0 = not optimistic and 10 = very optimistic). Ratings from all 8 weeks were averaged.
Time Frame: Week 1 of intervention - Week 8 of intervention
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Positive Psychology
Number analyzed (Participants) | 20
score on a scale
  pre-exercise | 8.0 (1.8)
  post-exercise | 8.6 (1.4)

10. Secondary Outcome: Immediate Impact of Exercises: Positive Affect Score
Description: Participants will provide ratings of their present level of positive affect after each PP exercise, measured on a 10-point Likert scale (score range: 0-10, 0 = not happy and 10 = very happy). Ratings from all 8 weeks were averaged.
Time Frame: Week 1 of intervention - Week 8 of intervention
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Positive Psychology
Number analyzed (Participants) | 20
score on a scale
  pre-exercise | 7.9 (1.6)
  post-exercise | 8.5 (1.5)

ADVERSE EVENTS:
Time Frame: 8 weeks
Arm/Group | Positive Psychology
All-Cause Mortality (participants affected / at risk) | 1/20
Serious Adverse Events (participants affected / at risk) | 1/20
Other Adverse Events (participants affected / at risk) | 0/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Positive Psychology (N=20)
Death due to complications related to hematopoietic stem cell transplantation (Blood and lymphatic system disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-08-09): https://cdn.clinicaltrials.gov/large-docs/04/NCT03654404/Prot_SAP_000.pdf